CLINICAL TRIAL: NCT02335502
Title: A Post Market Cohort to Assess the Performance of the Spinal Modulation Neurostimulator System for the Management of Chronic Intractable Pain
Brief Title: A Post Market Study to Assess the Spinal Modulation Neurostimulator System for Chronic Intractable Pain
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 04-SMI-2012
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Results first posted 2017-08-03 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treated Subjects: All subjects recruited and treated with the Axium neurostimulator
  Interventions: Device: Implantation with the commercially available Axium neurostimulator

INTERVENTIONS:
Device: Implantation with the commercially available Axium neurostimulator

SUMMARY:
04-SMI-2012 is post market, observational, questionnaire based study to assess the effectiveness of the commercially available Axium neurostimulator in the management of chronic, intractable pain.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old
2. Subject is able and willing to comply with the follow-up schedule and protocol
3. Chronic, intractable pain in the thoracic, lumbar and/or sacral distribution(s) for at least 6 months
4. Failed conservative treatments for chronic pain including but not limited to pharmacological therapy, physical therapy and interventional pain procedures for chronic pain
5. Minimum baseline pain rating of 60 mm on the Visual Analog Scale in the primary region of pain
6. In the opinion of the Investigator, the subject is psychologically appropriate for the implantation for an active implantable medical device
7. Subject is able to provide written informed consent
8. Subject speaks Dutch or English

Exclusion Criteria:

1. Female subject of childbearing potential is pregnant/nursing, plans to become pregnant or is unwilling to use approved birth control
2. Escalating or changing pain condition within the past month as evidenced by investigator examination
3. Subject has had corticosteroid therapy at an intended site of stimulation within the past 30 days
4. Subject has had radiofrequency treatment of an intended target Dorsal Root Ganglion within the past 3 months
5. Subject currently has an active implantable device including implantable cardioverter defibrillator, pacemaker, spinal cord stimulator or intrathecal drug pump
6. Patient has pain only or primarily within a cervical dermatomal distribution
7. Subject is unable to operate the device
8. Subjects with indwelling devices that may pose an increased risk of infection
9. Subjects currently has an active infection
10. Subject has, in the opinion of the Investigator, a medical comorbidity that contraindicates placement of an active medical device
11. Subject has participated in another clinical investigation within 30 days
12. Subject has a coagulation disorder or uses anticoagulants that, in the opinion of the investigator, precludes participation
13. Subject has been diagnosed with cancer in the past 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Pain Patients
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2012-04; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - St Antonius Ziekenhuis, Nieuwegein
  - Erasmus MC Pijnbehandelcentrum, Rotterdam

RESULTS

PARTICIPANT FLOW:
Groups:
- All Enrolled Subjects: All subjects enrolled into the study with intent to treat with the Axium Neurostimulator
Period: Overall Study
Arm/Group | All Enrolled Subjects
Started | 66
Received Trial System | 65
Receiving Permanent System | 56
Completed | 49
Not Completed | 17

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 66
Age, Continuous [Mean (Full Range); unit: years] | 52 [30 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 65
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 66

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity for Overall Pain From Pre-treatment Baseline
Description: The Visual Analog Scale (VAS) is self-administered instrument assessing average pain intensity. Subjects rated their pain on a horizontal line, 10 cm in length, anchored by word descriptors on each end (no pain to worst imaginable pain). A higher score indicates a higher pain level. The values range from 0 (minimum pain) to 10 (maximum pain).
Time Frame: 3, 6 and 12-Months
Population: Differences in participants over time is due to early withdrawals and missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Subjected Treated With the Permanent Implantable Axium System: All subjects treated with the Axium implantable neurostimulator
Arm/Group | Subjected Treated With the Permanent Implantable Axium System
Number analyzed (Participants) | 56
units on a scale
  Baseline | 7.4 (1.41)
  3-Months: number analyzed (Participants) | 48
  3-Months | 3.9 (2.63)
  6-Months: number analyzed (Participants) | 45
  6-Months | 4.5 (2.84)
  12-Months: number analyzed (Participants) | 49
  12-Months | 4.7 (2.87)

2. Primary Outcome: Percentage of Subjects With at Least 50% Pain Reduction
Description: Percent of subjects with at least a 50% reduction from the baseline pain VAS to the end of trial period VAS. The Visual Analog Scale (VAS) is self-administered instrument assessing average pain intensity. Subjects rated their pain on a horizontal line, 100 mm in length, anchored by word descriptors on each end (no pain to worst imaginable pain). A higher score indicates a higher pain level.
Time Frame: Baseline and End of Trial Visit
Population: All subjects treated with the Axium implantable neurostimulator who completed their end of trial visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjected Treated With the Permanent Implantable Axium System
Number analyzed (Participants) | 47
Participants
  >= 50% Pain Reduction | 29
  < 50% Pain Reduction | 18

ADVERSE EVENTS:
Time Frame: All adverse events reported spontaneously by the subject or observed by the investigator or his staff were recorded from the time of enrollment to study completion or early withdrawal.
Arm/Group | All Enrolled Subjects
Serious Adverse Events (participants affected / at risk) | 8/66
Other Adverse Events (participants affected / at risk) | 7/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=66)
Dural puncture (Injury, poisoning and procedural complications) | 1 (1)
Hematoma/Infection (Injury, poisoning and procedural complications) | 1 (1)
Infection (Infections and infestations) | 4 (4)
Motor deficit-transient (Injury, poisoning and procedural complications) | 1 (1)
Return of symptoms/worsening of disease state (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=66)
Hematoma (became SAE) (Injury, poisoning and procedural complications) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Infection (became SAE) (Infections and infestations) | 1 (1)
Loss of stimulation (Injury, poisoning and procedural complications) | 2 (2)
Pain at IPG site (Injury, poisoning and procedural complications) | 2 (2)
Spinal tap headache (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days